CLINICAL TRIAL: NCT06499025
Title: A Clinical Study to Evaluate the Safety and Initial Efficacy of Targeted AML1-ETO Neoantigen Cytotoxic T Cells (CTL) in the Treatment of Relapsed or Refractory t(8; 21) AML
Brief Title: Treatment of Relapsed or Refractory t(8; 21) AML With Targeted AML1-ETO Neoantigen Cytotoxic T Cells (CTL)
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: BGI, China (Other)
Collaborators: Shenzhen University General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGI-007; KYLLHS-20230402A (Other: Ethics Committee of Shenzhen University General Hospital)
Record Dates: First submitted 2024-07-07; First posted 2024-07-12 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: AML; t(8;21); Neoantigen
MeSH Terms: interventions — Cyclophosphamide; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- targeted AML1-ETO neoantigen cytotoxic T cells (CTL) (Experimental): The escalating doses of cells (CTL) in this study will be 5*10^7 cells and 1*10^8 cells.
  Interventions: Biological: targeted AML1-ETO neoantigen cytotoxic T cells (CTL); Drug: Cyclophosphamide injection; Drug: Decitabine Injection; Drug: Liposome mitoxantrone

INTERVENTIONS:
Biological: targeted AML1-ETO neoantigen cytotoxic T cells (CTL) — After subject screening, peripheral blood mononuclear cell #PBMC# donors matching half or more of the subject's HLA matching will undergo blood collection to prepare neoantigen cytotoxic T cells. Neoantigen cytotoxic T cells preparation is expected to be 25-30 days after blood collection. In this study, the bridging therapy will be allowed before Chemotherapy preconditioning. Chemotherapy preconditioning will be performed before neoantigen cytotoxic T cells transfusion.
Drug: Cyclophosphamide injection — Cyclophosphamide injection will be performed in -10 to -8d before neoantigen cytotoxic T cells transfusion
Drug: Decitabine Injection — Decitabine Injection will be performed in -12 to -8d before neoantigen cytotoxic T cells transfusion
Drug: Liposome mitoxantrone — Liposome mitoxantrone will be performed in -9 to -8d before neoantigen cytotoxic T cells transfusion

SUMMARY:
1. To evaluate the safety and tolerability of targeted AML1-ETO neoantigen cytotoxic T cells (CTL) in the treatment of relapsed or refractory acute myeloid leukemia .
2. To evaluate the effectiveness of targeted AML1-ETO neoantigen cytotoxic T cells (CTL)，by the complete response rate(CRR) and overall survival (OS) followed.

DETAILED DESCRIPTION:
This is a single arm、open label and non-randomied clinical trial ，divided into dose exploration phase (Part A) and dose extension phase (Part B).

Part A: Plan to enroll six subjects to evaluate the safety and tolerabilty of targeted neoantigen cytotoxic T cells (CTL),determine dose-limiting toxicity(DLT),explore the maximum tolerated dose (MTD) or the recommended dose for later clilnical studies.The DLT observation period is 28 days after the infusion of targeted neoantigen cytotoxic T cells (CTL) iniection. One dose group(total number of cells is 5×10^7/bag) and the another one (total number of cells is 10×10^7 /bag )is setted by the 3+3 test design.

Part B: Ten subjects are planned to be enrolled in the dose-exploration phase with the recommended dose, to further evaluate the safety、tolerability and its efficacy of targeted neoantigen cytotoxic T cells (CTL) in relapsed or refractory acute myeloid leukemia.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old (including 18, 75 years old), gender is not limited;
2. According to WHO (2020) criteria, the subjects are diagnosed for recurrent or refractory t(8:21) acute myeloid leukemia or demonstrated persistant AML1-ETO positiving or genetic MRD recurrence after ≥3 cycles of intensive chemotherapy, as confirmed by quantitative PCR;
3. The subjects voluntarily participate in the study and sign the Informed Consent Form by themselves or their legal guardians;
4. The HLA types of subjects are HLA-A* 11:01 or HLA-A*02:01;
5. Possessing the AML1-ETO(RUNX1-RUNX1T1) funsion gene;
6. Disease progression after adequate first-line systemic treatment for remission, or disease progression after first-line or above systemic systemic treatment for ≥2 cycles , or without remission (CR or PR) after≥4 cycles of treatment ;
7. No contraindications for collection of mononuclear cells from peripheral blood ;
8. ECOG score ≤1;
9. The survival time is exspected to be≥ 3 months;
10. Have the ability to understand and be willing to sign the informed consent for this test.

Exclusion Criteria:

1. Tumor cells do not express AML1-ETO neoantigen;
2. Active infection;
3. Abnormal liver function [TBil（total bilirubin)>1.5×ULN, ALT>2.5×ULN], abnormal kidney function [Scr（serum creatinine)>1.5×ULN];
4. Unstable angina or 3/4 class of congestive heart failure according to New York Heart Association, or multiple organ dysfunction;
5. HIV/AIDS patients;
6. Participants who need treatment of long-term anticoagulation (warfarin or heparin) or antiplatelet(aspirin>300mg/d; Clopidogrel>75mg/d) ;
7. Participants who received radiotherapy within 4 weeks ,prior to study initiation (blood collection);
8. Known or suspected drug abuse or alcohol dependence;
9. Patients with mental disorders or other medical conditions are unable to obtain informed consent and cooperate to complete the requirements of experimental treatment and examination procedures;
10. Participants in other clinical trials within 30 days;
11. Pregnant or lactating women and male subjects (or their partners) or female subjects who plan to become pregnant during the study period and within 6 months after the end of the study ,and do not wish to use a medically approved effective contraceptive method (such as an IUD or condom) during the study period;
12. The investigator evaluates that the subject is unable or unwilling to comply with the requirements of the study protocol;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety assessment (Evaluation of treatment-related adverse events according to CTCAEv5.0) | From preconditioning or cell reinfusion to one year after cell reinfusion or the initiation of other antitumor therapy or the discontinuation of the trial for other reasons, whichever occurred first.
  To determine the incidence of AE and SAE in clinical trials

SECONDARY OUTCOMES:
Complete response rate | Up to 48 weeks
  The total number of subjects with complete response (CR) confirmed and the proportion of subjects in the corresponding analysis set
Overall survival (OS) | Up to 72 weeks
  The time from cell transfusion to death who have completed the prescribed dose. If the sujects is lost to follow-up, the last known date of surival wil be OS deletion time

CONTACTS AND LOCATIONS:
Overall Officials: LiXin Wang, Doctor, Principal Investigator — Shenzhen University General Hospital
Locations (1):
- Shenzhen University General Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Godugu K, Rajabi M, Mousa SA. RETRACTED: Godugu et al. Anti-Cancer Activities of Thyrointegrin alphavbeta3 Antagonist Mono- and Bis-Triazole Tetraiodothyroacetic Acid Conjugated via Polyethylene Glycols in Glioblastoma. Cancers 2021, 13, 2780. Cancers (Basel). 2024 May 15;16(10):1880. doi: 10.3390/cancers16101880. PMID 38792024
- [Background] Falini B, Mecucci C, Tiacci E, Alcalay M, Rosati R, Pasqualucci L, La Starza R, Diverio D, Colombo E, Santucci A, Bigerna B, Pacini R, Pucciarini A, Liso A, Vignetti M, Fazi P, Meani N, Pettirossi V, Saglio G, Mandelli F, Lo-Coco F, Pelicci PG, Martelli MF; GIMEMA Acute Leukemia Working Party. Cytoplasmic nucleophosmin in acute myelogenous leukemia with a normal karyotype. N Engl J Med. 2005 Jan 20;352(3):254-66. doi: 10.1056/NEJMoa041974. PMID 15659725
- [Background] Biernacki MA, Foster KA, Woodward KB, Coon ME, Cummings C, Cunningham TM, Dossa RG, Brault M, Stokke J, Olsen TM, Gardner K, Estey E, Meshinchi S, Rongvaux A, Bleakley M. CBFB-MYH11 fusion neoantigen enables T cell recognition and killing of acute myeloid leukemia. J Clin Invest. 2020 Oct 1;130(10):5127-5141. doi: 10.1172/JCI137723. PMID 32831296
- [Background] Blankenstein T, Leisegang M, Uckert W, Schreiber H. Targeting cancer-specific mutations by T cell receptor gene therapy. Curr Opin Immunol. 2015 Apr;33:112-9. doi: 10.1016/j.coi.2015.02.005. Epub 2015 Feb 27. PMID 25728991
- [Background] Sahin U, Tureci O. Personalized vaccines for cancer immunotherapy. Science. 2018 Mar 23;359(6382):1355-1360. doi: 10.1126/science.aar7112. PMID 29567706
- [Background] van der Lee DI, Reijmers RM, Honders MW, Hagedoorn RS, de Jong RC, Kester MG, van der Steen DM, de Ru AH, Kweekel C, Bijen HM, Jedema I, Veelken H, van Veelen PA, Heemskerk MH, Falkenburg JHF, Griffioen M. Mutated nucleophosmin 1 as immunotherapy target in acute myeloid leukemia. J Clin Invest. 2019 Feb 1;129(2):774-785. doi: 10.1172/JCI97482. Epub 2019 Jan 14. PMID 30640174